CLINICAL TRIAL: NCT02021110
Title: An International, Multicenter, Randomized Controlled Clinical Trial Assessing the Efficacy of Ursodeoxycholic Acid as a Volume Reducing Treatment in Symptomatic Polycystic Liver Disease
Brief Title: Ursodeoxycholic Acid as Treatment for Polycystic Liver Disease
Acronym: CURSOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLD 11-01
Record Dates: First submitted 2013-12-12; First posted 2013-12-27 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2016-04

CONDITIONS: Polycystic Liver Disease; Polycystic Kidney, Autosomal Dominant
MeSH Terms: conditions — Polycystic liver disease; Polycystic Kidney, Autosomal Dominant | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): This group will receive standard care (no treatment)
- Ursodeoxycholic Acid (Experimental): The intervention group will receive 15-20mg/kg/day UDCA for 24 weeks
  Interventions: Drug: Ursodeoxycholic Acid

INTERVENTIONS:
Drug: Ursodeoxycholic Acid — The intervention group will receive 15-20mg/kg/day UDCA for 24 weeks
  Other Names: Ursochol
  Arms: Ursodeoxycholic Acid

SUMMARY:
Rationale: Polycystic liver disease (PLD) is a rare disorder characterized by >20 fluid-filled hepatic cysts. Polycystic livers are present in the combination with renal cysts as a manifestation of autosomal dominant polycystic kidney disease (ADPKD), or isolated in the absence of renal cysts as autosomal dominant polycystic liver disease (ADPLD or PCLD). PLD patients are confronted with symptoms caused by the mass effect of their polycystic liver every day for the rest of their life. There is no standard therapeutic option for symptomatic PLD patients. Current options are fairly invasive or their efficacy is only moderate.

Preliminary data in our research lab have shown that ursodeoxycholic acid (UDCA) inhibited the proliferation of polycystic human cholangiocytes in vitro through the normalization of the intracellular calcium levels in cystic cholangiocytes. The investigators also found that daily oral administration of UDCA for 5 months to polycystic kidney disease (PCK) rats, an animal model of ARPKD that spontaneously develops hepato-renal cystogenesis, resulted in inhibition of hepatic cystogenesis.

The investigators hypothesize that UDCA is an effective therapeutic tool in reducing liver volume in PLD.

Objective: First, to demonstrate whether UDCA-therapy is effective in reducing total liver volume in PLD patients. Second, the investigators want to assess if UDCA modifies quality of life. Finally, the investigators want to assess safety and tolerability.

Study design: International, multicenter, randomized, controlled trial Study population: 34 subjects (18 ≤age ≤ 80 years) suffering from symptomatic polycystic liver disease with underlying diagnosis of (PCLD or ADPKD), defined as ≥ 20 liver cysts on CT-scan and liver volume of ≥ 2500. Symptomatic is defined as Eastern Cooperative Oncology Group- Performance Score (ECOG-PS) ≥ 1 and having at least three out of ten PLD symptoms.

Intervention: The patients will be randomized (1:1) into two groups. One group of patients will receive 15-20mg/kg/day UDCA for 24 weeks. The other group will receive standard care.

Main study endpoint: Proportional change of total liver volume in UDCA treated patients versus non treated patients, as assessed by CT at baseline and 6 months.

DETAILED DESCRIPTION:
We investigated whether ursodeoxycholic acid was able to reduce total liver volume in polycystic liver disease.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ age ≤ 80 years
* Polycystic liver disease with underlying diagnosis of (PCLD or ADPKD), defined as ≥ 20 liver cysts
* Total liver volume ≥ 2500 mL
* Symptomatic defined as ECOG-PS ≥ 1 (2), and having at least three out of ten PCLD symptoms:
* Informed consent, patients are willing and able to comply with the study drug regimen and all other study requirements.

Exclusion Criteria:

* Use of oral anticonceptives or estrogen supplementation
* Use of UDCA in 3 months before baseline
* Females who are pregnant or breast-feeding or patients of reproductive potential not employing an effective method of birth control.
* Intervention (aspiration or surgical intervention) within six months before baseline
* Treatment with somatostatin analogues within six months before baseline
* Renal dysfunction (MDRD-Glomerular filtration rate< 30 ml/min/1.73m2)
* Patients with a kidney transplant
* Hypersensitivity reaction to UDCA or patients with galactose-intolerance, lactase deficiency or glucose-galactose malabsorption
* Acute cholecystitis or frequent biliary colic attacks
* Acute stomach or duodenal ulcers
* Inflammation of small intestine or colon
* Use of drugs that can interact with UDCA, such as colestyramine, aluminium hydroxide or cyclosporin
* Enrolment in another clinical trial of an investigational agent while participating in this study
* History or other evidence of severe illness or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* Mental illness that interferes with the patient ability to comply with the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Effect of UDCA on total liver volume | Baseline to week 24
  Proportional change of total liver volume in UDCA treated patients versus non treated patients, as assessed by CT at baseline and week 24

SECONDARY OUTCOMES:
Effect of UDCA-therapy on absolute total liver volume | Baseline to week 24
  Absolute total liver volume at baseline and end of treatment (week 24) will be measured
Effect of UDCA on gastro-intestinal symptoms measured by a GI-questionnaire | Baseline to week 24
  Improvement in Gastrointestinal Symptom score
Effect of UDCA on health related quality of life as measured by Study Form -36 | Baseline to week 24
  Improvement in Study Form -36 score
Proportion of patients with any reduction in total liver volume after 24 weeks | Baseline to week 24
  Proportion reduction in total liver volume
Effect of UDCA on absolute total kidney volume | Baseline to week 24
  Change in total kidney volume after 24 weeks

OTHER OUTCOMES:
Adverse events as a measure of tolerability and safety of UDCA | Baseline to week 24
  All adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Joost PH Drenth, dr., Principal Investigator — Radboud University Medical Centre Nijmegen, the Netherlands
Locations (3):
- Netherlands (2):
  - Radboud University Medical Centre Nijmegen, Nijmegen, Gelderland
  - Academic Medical Centre Amsterdam, Amsterdam
- Donostia University Hospital, Donostia / San Sebastian, Spain

REFERENCES:
- [Derived] D'Agnolo HM, Kievit W, Takkenberg RB, Riano I, Bujanda L, Neijenhuis MK, Brunenberg EJ, Beuers U, Banales JM, Drenth JP. Ursodeoxycholic acid in advanced polycystic liver disease: A phase 2 multicenter randomized controlled trial. J Hepatol. 2016 Sep;65(3):601-7. doi: 10.1016/j.jhep.2016.05.009. Epub 2016 May 17. PMID 27212247